CLINICAL TRIAL: NCT00348270
Title: Comparison of the Quality of Vision Provided by AMO Tecnis Z9000 Three-piece Silicone Posterior Chamber Intraocular Lens and Alcon Laboratories MA60 Acrysof Three-piece Acrylic Posterior Chamber Intraocular Lens
Brief Title: Comparison of the Quality of Vision Provided by AMO Tecnis Z9000 and Alcon Laboratories MA60 Acrysof Posterior Chamber Intraocular Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R367/25/2004
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Cataract
Keywords: Cataract; Intraocular lens; Aberration; Wavefront
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Device: Tecnis Z9000 intraocular lens
Device: MA60 intraocular lens

SUMMARY:
This study is a comparison of the quality of vision provided by AMO Tecnis Z9000 three-piece silicone posterior chamber intraocular lens and Alcon Laboratories MA60 three-piece acrylic posterior chamber intraocular lens.

DETAILED DESCRIPTION:
Today, intraocular lenses (IOLs) are routinely implanted after cataract extraction. Cataract surgical techniques are constantly developing due to innovations in surgical implantation and IOL manufacturing processes. Although material development and surgical implantation have advanced extensively during the past several years, there has been little attention paid to the improvement of the optical quality of IOLs.

It has been documented that the vision of an IOL patient is no better than that of a person with healthy eyes of a similar age, i.e., when a 65-year-old patient with cataracts has them removed and implanted with an IOL, the resulting visual outcome is no better than the visual quality of a 65-year-old without cataracts. The fact that the visual quality of the IOL patients is no better than that of their same-age counterparts is surprising because an IOL is optically superior to the natural crystalline lens. This fact may be explained by aberrations.

Aberrations cause incoming light that would otherwise be focused to a point to be blurred, which in turn causes a reduction in visual quality. This reduction in quality is more severe under low luminance conditions because ocular aberrations increase when the pupil size gets larger. The Z9000 is an IOL that is designed to counteract the spherical aberration of the cornea and thus improve the resulting visual quality of IOL patients.

Different materials and lens designs result in different visual quality. The handling of the lens, proper centration in the eye, the postoperative course, and the optical image may vary depending on the design of the lens. Two lenses will be compared: AMO Tecnis Z9000 three-piece silicone lens and Alcon Laboratories MA60 three-piece acrylic lens.

This will be a randomized, evaluator-masked study in bilateral cataract surgery patients. Each patient will be assigned to a AMO Tecnis Z9000 lens in one eye and an Alcon Laboratories MA60 lens in the other eye. All first surgeries will be on the right eye. A randomization list will be used to decide lens allocation.

A total of 80 patients (men and women) from the Singapore National Eye Centre will be enrolled in the study. All patients will undergo wavefront analysis 90-120 days postoperatively.

The two lens models look different, even in the eye, after implantation. It is not possible to mask the individual investigator at the time of surgery or personnel responsible for conducting the clinical ocular examinations (e.g., evaluation of complications, posterior capsule, IOP, pupil size) and optic evaluations (e.g., evaluation of the IOL).

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral cataracts, eligible for phacoemulsification with primary implantation of a posterior chamber IOL
2. Males and females 50 to 80 years of age
3. Expected maximum of 6-weeks and minimum of 3 weeks interval between a single patient's surgeries
4. Best corrected visual acuity (BCVA) should be no better than 20/40 in the presence of a glare source. (In the early treatment diabetic retinopathy study [ETDRS] visual acuity chart, better than 20/40 will be at least 3 letters read correctly in the 20/30 line).
5. Best corrected visual acuity projected by Potential Acuity Meter (PAM) or other reliable potential acuity test procedure to be 20/30 or better in each eye after cataract removal and IOL implantation.
6. Naturally dilated pupil size (in dim light) ≥ 4.0 mm (with no dilation medications) - both eyes
7. Anticipated correction with an IOL of +6 to +30 diopters (both eyes)
8. Evidence of a personally signed and dated informed consent document indicating the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the trial
9. Willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

1. Preoperative pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmus or macrophthalmus, optic nerve atrophy
2. Previous intraocular or corneal surgery, including refractive surgery, corneal transplant
3. Other pathologies potentially affecting visual acuity, e.g., macular degeneration, glaucoma with the presence of visual field defects
4. An increased risk for complications which could require vitreoretinal surgery
5. Corneal irregularities potentially affecting visual acuity, e.g., keratoconus, corneal dystrophy
6. Corneal opacities
7. Keratometric astigmatism exceeding 1.5 diopters
8. Patient in whom postoperative refractive error is planned to be different between fellow eyes (anisometropia) such as in cases where postoperative refraction is planned for mono-vision
9. Current contact lens usage (within 6 months prior to first surgery and/or during the study)
10. Other ocular surgery at time of cataract extraction
11. Uncontrolled diabetes
12. Any neurological condition that might interfere with performance of required tests
13. Immune deficiency disease
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
15. Use of any systemic or topical drug known to interfere with visual performance

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this comparative study is the best corrected mesopic log contrast sensitivity function of eyes implanted with Z9000 and MA60 lenses at 6 cycles/degree, 90-120 days postoperatively.

SECONDARY OUTCOMES:
The best corrected mesopic log contrast sensitivity function of eyes implanted with Z9000 and MA60 lenses at 1.5, 3, 12, and 18 cycles/degree, 90-120 days postoperatively
The change in best corrected mesopic log contrast sensitivity function after cataract surgery (postoperatively minus preoperatively) at 1.5, 3, 6, 12, and 18 cycles/degree
The residual spherical aberrations of the postoperative eye using wavefront analysis
Logarithm of the minimum angle of resolution (LogMAR) visual acuity
Postoperative ocular complications/adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Han Chua, Principal Investigator — Singapore National Eye Center
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore